CLINICAL TRIAL: NCT01236989
Title: Anatomical Liver Resection by Means of Ultrasound-guided Vessel Compression Versus Non-anatomical Resection for Hepatocellular Carcinoma: A Randomized Controlled Trial
Brief Title: Prognostic Impact of Anatomical Resection Vs. Non-anatomical Resection for HCC
Acronym: ARversusNAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Responsible Party: Guido Torzilli, MD, PhD, Liver Surgery Unit, 3rd Department of Surgery, University of Milan School of Medicine, IRCCS Istituto Clinico Humanitas, Rozzano, Milan, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR vs NAR
Record Dates: First submitted 2010-10-29; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-10

CONDITIONS: Patients Affected by Hepatocellular Carcinoma; Disease-Free Survival; Overall Survival
Keywords: anatomical resection; non-anatomical resection; IOUS-guided finger compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anatomical resection (Experimental)
  Interventions: Procedure: anatomical liver resection
- Non-anatomical resection (Active Comparator)
  Interventions: Procedure: Non-anatomical liver resection

INTERVENTIONS:
Procedure: anatomical liver resection — anatomical liver resection by means of IOUS-finger compression
  Arms: Anatomical resection
Procedure: Non-anatomical liver resection — non-anatomical liver resection
  Arms: Non-anatomical resection

SUMMARY:
Prognostic impact of AR vs NAR

DETAILED DESCRIPTION:
Whether anatomical is better than non anatomical resection for HCC is still debated. This prospective randomized study aimed to address which approach is better in terms of patients prognosis.

ELIGIBILITY:
Inclusion Criteria:

* patient affected by single HCC
* patients in whom liver resection is indicated
* HCC without vascular invasion and/or thrombosis

Exclusion Criteria:

* multinodular HCC
* metastatic disease
* spontaneous tumor rupture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the prognostic impact of anatomical resection by means of intraoperative ultrasound (IOUS) guided vessel compression versus nonanatomical resection in terms of disease free and overall survival | 5-years

SECONDARY OUTCOMES:
the impact of anatomical resection versus non-anatomical resection in terms of postoperative mortality and morbility | 30 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Principal Investigator — IRCCS Istituto Clinico Humanitas, Milan, Italy
Locations (1):
- IRCCS Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Background] Hasegawa K, Kokudo N, Imamura H, Matsuyama Y, Aoki T, Minagawa M, Sano K, Sugawara Y, Takayama T, Makuuchi M. Prognostic impact of anatomic resection for hepatocellular carcinoma. Ann Surg. 2005 Aug;242(2):252-9. doi: 10.1097/01.sla.0000171307.37401.db. PMID 16041216
- [Background] Torzilli G, Procopio F, Cimino M, Del Fabbro D, Palmisano A, Donadon M, Montorsi M. Anatomical segmental and subsegmental resection of the liver for hepatocellular carcinoma: a new approach by means of ultrasound-guided vessel compression. Ann Surg. 2010 Feb;251(2):229-35. doi: 10.1097/SLA.0b013e3181b7fdcd. PMID 19838106
- [Background] Torzilli G, Makuuchi M. Ultrasound-guided finger compression in liver subsegmentectomy for hepatocellular carcinoma. Surg Endosc. 2004 Jan;18(1):136-9. doi: 10.1007/s00464-003-9024-x. Epub 2003 Nov 21. PMID 14625736